CLINICAL TRIAL: NCT04263857
Title: Register of Survey and Evaluation of Blood Stem Cell Transplantations of Clinic III of Internal Medicine III
Brief Title: Register of Blood Stem Cell Transplantation
Acronym: REBB3M
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: REBB3M
Record Dates: First submitted 2018-03-02; First posted 2020-02-11 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancies
Keywords: autologous & allogenic blood stem cell transplantations
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Register of patients with blood stem cell transplantations (autologous, allogen).

DETAILED DESCRIPTION:
Documenting the success rate in terms of complication rate, disease response, survival rate, engraftment, and details of transplantation settings, for example donor and conditioning data, remission status before transplantation.

It's a register of patients who have one or more autologous and / or allogenic blood stem cell transplants due to an existing indication for performing myeloablative / non-myeloablative high-dose chemotherapy.

The inclusion occurs at our center during preparation for blood stem cell transplantation. The written consent will be obtained separately in the context of the information on blood stem cell transplantation. Participation is voluntary and consent can be revoked at any time. This involves no additional effort for the patient and has no influence on his treatment. It may be necessary in the course of contacting the patient at home, as long as the data is incomplete. This is also explicitly explained. A copy of the declaration of consent is given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* signed IC
* patients eligible for stem cell transplantation

Exclusion Criteria:

* unable to consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults, Age >= 18 years
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2037-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
Register of stem cell transplantation | approximately over 20 years
  Recording of all stem cell transplantations over many years

SECONDARY OUTCOMES:
Register of toxicities | approximately over 20 years
  Recording of toxicities occured during and after SCT according to GvHD Score Standards and blood and bone marrow samples, and Imaging (CT Scans)
Register of complications | approximately over 20 years
  Recording of complications occurred during and after SCT in Terms of infectious complications and occurance of GvHD (according to GvHD Score and Imaging and clinical assessment)
Register of morbidities | approximately over 20 years
Register of survivals | approximately over 20 years
  Recording of survival Status, Assessment of Remission Status by bone marrow and blood diagnostics, clinical follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mareike Verbeek, MD, Principal Investigator — Klinikum rechts der Isar der TU Munich, Germany
Locations (1):
- Klinikum rechts der Isar der TU München, Munich, Germany

IPD SHARING:
Plan to Share IPD: No